CLINICAL TRIAL: NCT03199222
Title: Prosthetic Smart Socket Technology to Improve Patient Interaction, Usability, Comfort, Fit, and Function.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Collaborators: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00026455
Record Dates: First submitted 2017-04-04; First posted 2017-06-26 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Complications of the Amputated Limb
Keywords: amputation; transtibial; socket; pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Smart socket technology w/patient prompting (Experimental): The prosthetic user WILL receive prompting by the smart socket technology regarding improper fit and suggestions for how to a restore a proper fit (i.e socks). Investigators will have access to the Smart Socket Technology database.
  Interventions: Device: Prosthetic smart socket technology with patient prompting
- Arm 2: Clinical protocol. No patient prompting (No Intervention): The prosthetic user WILL NOT receive prompting by the smart socket technology regarding improper fit and suggestions for how to a restore a proper fit (i.e socks). However, investigators will have access to the Smart Socket Technology database.

INTERVENTIONS:
Device: Prosthetic smart socket technology with patient prompting — The smart socket technology will send feedback to the user's smartphone with suggestions including the removal or application of prosthetic socks over the residual limb or other volume management strategies to improve fit and comfort.
  Arms: Arm 1: Smart socket technology w/patient prompting

SUMMARY:
A common problem for the intermediate preparatory stage of prosthetic rehabilitation is distal pressure, due to commonly compromised sensation and lack of understanding how to address it in a newly fitted prosthesis. Excessive pressure can lead to severe skin breakdown, infection, surgical revision, re-hospitalization and delayed rehab. To prevent this common problem among rehabilitating amputees, smart socket technology has been developed to better identify problems that may occur. The Smart Socket Technology including Prompting (SST+P) in this pre-clinical project proposal provides a step activity monitor and senses distal pressure, which is novel to the technology. When excessive pressure is sensed on the residual limb, it will send a signal to the user's smart phone to make an adjustment. This prompting improves patient interaction and may prevent problems as a result of common volume fluctuation and compromised sensation. The purpose of this clinical trial is to determine if the ALPS iForce smart socket technology with prompting (SST+P) will improve patient interaction, usability, comfort, fit, function and health economy outcomes compared with the standard of care (SOC) clinical practice protocols of fitting prosthetic socket interfaces

DETAILED DESCRIPTION:
Limb loss requires prosthetic use. Prostheses usually consist of 2 components: 1) a soft interface to protect the skin and underlying musculoskeletal tissue and 2) a structural interface to enable attachment of prosthetic components to the human body. The interface connects the patient's body to the prosthetic components and thus ground during gait. The interface has 2 purposes: 1) to distribute weight-bearing forces throughout the entire residual limb (RL) and 2) to suspend the prosthesis during swing phase and unweighting. The interface assists in distributing vertical loads during weight bearing to minimize focal loading on pressure intolerant tissues. The interface also suspends prosthetic components to the RL in swing phase and other periods of unweighting.

Many amputees experience RL complications and decreased mobility resulting from the inability to detect excess pressure or a lack of distal contact with newly fit and poorly fit interfaces. A smart socket technology interface could benefit every new prosthetic patient by prompting the user of a compromised socket fit prior to inhibiting functional use and safety. Further, the smart socket technology interface may ultimately prevent other health complications and improve patient interaction, usability, comfort, fit and function. The ALPS iForce most economically measures these variables more comprehensively than any other known single device. Therefore the smart socket interface technology chosen for this proposal is the ALPs iForce. The iForce tracks pressure over time and indicates to the user when positive or negative distal pressure exists by providing volume management suggestions (i.e. sock-ply adjustments). The user interacts with data measured sent wirelessly to an application on a smart phone (Android/iOS/Windows), handheld device, or PC. Suggestions may include removal or application of prosthetic socks over the RL, or other appropriate volume management strategies, to improve fit and comfort. Early warning to possible skin irritation and breakdown may lead to a healthier limb.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral transtibial amputation
2. Unilateral revision or reconstruction of transtibial amputation
3. Candidate for intermediate stage (i.e. preparatory) socket fitting
4. Male or female, of any ethnicity
5. 18-60 yrs of age (i.e. active military age)
6. 100-275 lbs.

Exclusion Criteria:

1. Body weight <100 or >275 lbs
2. Does not speak English or Spanish
3. Any other level of amputation than unilateral TTA

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-03-29 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Intermediate stage prosthetic complications | Will be tracked for 120 days.
  Clinical documentation will track incidence of dermatologic issues, skin breakdown, sock ply, circumference, infection and wound severity.
Limb volume activity of the residual limb | Will be tracked for 120 days
  Limb volume will be tracked through clinical documentation including residual limb volumetrics (circumferential measurements), sock-ply changes (journal), and required interface changes will be used to record volume activity and corresponding consequence and management strategies.
Intermediate stage prosthetic complications (clinical documentation) | Will be tracked for 120 days
  Re-hospitalization rate
Intermediate stage prosthetic complications (clinical documentation) | Will be tracked for 120 days
  Revision rate will be documented

SECONDARY OUTCOMES:
Balance and Stability | 30 days post-amputation and at end of trial (120 days)
  Post-amputation balance and stability will be tested with the Amputee Mobility Predictor (AMP). The AMP is a brief physical assessment (≈15min to administer) to objectively determine a lower extremity amputee's functional level. Subjects are assessed by progressing through a hierarchy of mobility tasks including sitting balance, standing balance, obstacle crossing, variable gait speed and stair gait.
Mobility | 30 days post-amputation and at end of trial (120 days)
  L-Test of Functional Mobility and the 2 minute walk test will be used to assess mobility. The L-Test is practical in design and intended to be used in a standard clinical hallway.29 Subjects begins the test seated in a chair.
  The patient rises from the chair, walks three meters, turns 90 degrees and then walks an additional seven meters. Upon completing seven meters, the subject turns 180 degrees, returns, turns 90 degrees to face the chair, and returns the three meters to his chair, where they retake the seat.
Step Activity | 120 days
  The Smart Socket Technology in this proposal has the capability of measuring step count activity. Step activity monitoring is utilized to count the number of steps taken.
Step Activity | 120 days
  Step activity monitoring is used to count the duration of step bout activity per stepping episode.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Highsmith, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No